CLINICAL TRIAL: NCT02194127
Title: Efficacy and Tolerability of a Treatment Over 28 Days With a Bilberry Extract Standardised to a Content of 25% Anthocyanidines in Volunteers With Impaired Twilight and Night Vision
Brief Title: Efficacy and Tolerability of a Bilberry Extract in Volunteers With Impaired Twilight and Night Vision
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1147.2
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Anthocyan capsules (Experimental): capsules containing 160 mg standardised bilberry extract (25% anthocyanidines)
  Interventions: Drug: Anthocyan capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anthocyan capsules
  Arms: Anthocyan capsules
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to determine the efficacy of Anthocyan to improve impaired twilight and night vision and to test its tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (volunteers) with age-related impaired twilight and night
* Age 50 to 70, men or women
* Written informed consent
* Full visual acuity (vision ≥ 0.7) according to DIN Standard condition
* Refraction ≤ +/-6.0 in the highest main step
* Age-related findings in the ophthalmologic examination (anterior chamber and eye ground)
* Normal intraocular pressure (10-20 mmHg)

Exclusion Criteria:

* Diabetes mellitus
* Epilepsy
* Abnormal visual acuity or eye ground (e.g. clouding of the lens)
* Age related vision problems
* Glaucoma and macular degeneration
* Disease of the retina
* Consumption of anthocyan preparations during the past six months
* Opthalmologic pathology: cataract, visus < 0.7, retinal pathology, maculopathy, intraocular pressure (> 21 mmHg), known acute or chronic eye disease, use of hard contact lenses, eye surgery performed within the last 12 months
* Any serious disorder that might interfere with his/her participation in this study and the evaluation of the efficacy or safety of the test drug: e.g. diabetes mellitus, anamnestic indications of diabetic microangiopathy or polyneuropathy, renal insufficiency, hepatic or metabolic dysfunction, cardiovascular disease (hypertension > 160/100 mmHg), psychiatric disorder, myasthenia gravis, delirious state, albino
* Any treatment that might interfere with the evaluation of the test drug, in particular drugs with known influence on eye sight or adaptation (e.g. chloroquine, digitalis, ethambutol, chlorpromazine or phenothiazine derivatives such as thioridazine, periciazine, perphenazine)
* Known hypersensitivity to any of the ingredients of the study drug
* Drug and alcohol abuse
* Pregnancy, lactation, women of childbearing potential who do not use an established contraceptive
* Participation in another trial within the past 30 days

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 1998-11; Primary Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the maximum velocity of dilatation of the pupil | day 29

SECONDARY OUTCOMES:
Measurement of the maximum velocity of dilatation of the pupil | Days 1 and 8
Measurement of the initial pupil diameter | days 1, 8 and 29
Measurement of the latency time | Days 1, 8 and 29
Measurement of the absolute and relative constriction amplitude | Days 1, 8 and 29
Measurement of maximum velocity of contraction | Days 1, 8 and 29
Measurement of velocity of contraction 2 | Days 1, 8 and 29
Measurement of initial minimal contrast level | Days 1, 8 and 29
  Determined with Gecko Contrast card
Time to regain contrast vision at one level above the initial minimal contrast | days 1, 8 and 29
  Determined with Gecko Contrast card
Measurement of contrast threshold level at illumination 0.1 cd/m2 with glare | Days 1, 8 and 29
  determined with Mesoptometer II
Measurement of contrast threshold level at illumination 0.032 cd/m2 without glare | Days 1, 8 and 29
  determined with Mesoptometer II
Recovery time after dazzling | Days 1, 8 and 29
Change of potential (µVolt) in retina due to photo activation | Baseline, days 1, 8 and 29
  Measured with Standard Electroretinography (ERG)
Assessment of subjective efficacy based on a visual analogue scale (VAS) rating questionnaire | Pre-dose and days 1, 8 and 29
Assessment of clinical global impression on a 5-point rating scale | Day 29
Number of patients with adverse events | up to day 29
Number of patients with significant changes in laboratory parameters | Baseline and day 29